CLINICAL TRIAL: NCT01710774
Title: Effect of Telemedicine Follow-up Care in Primary Health Care Versus Traditional Follow-up in Specialist Health Care on the Healing Time for Diabetes-related Foot Ulcers - a Cluster-randomized Controlled Trial
Brief Title: Telemedicine Follow-up in Primary Health Care for Diabetes-related Foot Ulcers
Acronym: DiaFOTo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); Norwegian Diabetes Association (Other); Bergen University College (Other); The Research Council of Norway (Other); Norwegian Nurses Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUS-ID210
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Foot; Foot Ulcer
Keywords: Diabetic Foot; Diabetes Mellitus; Foot Ulcer; Wound Healing; Delivery of Health Care; Depression; sequela; Sick Leave; Quality of Life; Amputation; Legg ulcer; Hospitalization; Health Economics
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Diabetes Mellitus; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional follow-up (No Intervention): Traditional follow-up with standard consultations at the Section of Endocrinology. For some patients, this will include follow-up from nurses in the home care or general practice office related to wound care. However, this is not the standard procedure and will not take place in combination with telemedicine follow-up.
- Telemedicine follow-up care (Active Comparator): Telemedicine follow-up care for people with diabetes-related foot ulcers in municipal primary health care in collaboration with specialist health care
  Interventions: Procedure: Telemedicine follow-up care

INTERVENTIONS:
Procedure: Telemedicine follow-up care — Telemedicine follow-up care for people with diabetes-related foot ulcers in municipal primary health care in collaboration with specialist health care
  Arms: Telemedicine follow-up care

SUMMARY:
This study will investigate whether telemedicine follow-up care for people with diabetes-related foot ulcers and people with leg ulcers (without diabetes) in municipal primary health care in collaboration with specialist health care is an equivalent alternative to traditional outpatient clinical follow-up in specialist health care (noninferiority trial) in relation to healing time.

DETAILED DESCRIPTION:
The increasing prevalence of diabetes, especially type 2 diabetes, combined with a steadily increasing proportion of older people in the population, will present enormous challenges for health care services and the individual with diabetes in Norway. Therefore, health care services need to rapidly begin treatment for people with diabetes-related foot ulcers to ensure high-quality treatment.

Telemedicine innovations for health care services have developed considerably in recent decades. The National Health Plan for Norway (2007-2010) emphasizes that the use of information and communication technologies is an important way of achieving health policy aims in establishing more integrated diagnosis, treatment and care pathways across organizational boundaries. Qualitative studies of diabetes-related foot ulcers have shown that using telemedicine equipment enables follow-up care of similar quality to traditional consultations while enabling more flexible organization and greater patient satisfaction. A few minor quantitative studies show positive gains when telemedicine equipment is used in following up diabetes-related foot ulcers, but no randomized controlled studies have been performed in this field. Further, studies focusing on the more long-term effects are lacking.

The project is in accordance with national guidelines and will contribute to increasing the focus on research related to integrated care. The investigators expect this project to provide evidence about alternative care pathways with a holistic approach that could moderate increases in the cost of health care services by delivering a larger proportion of services in municipal primary care. The project will be able to provide new evidence on meeting the challenges of diabetes-related care more systematically and proactively. The investigators expect that the results of this study will contribute to showing the extent to which treatment at the lowest effective service level will be more cost-effective and of good or better quality than traditional clinical follow-up. This study can and will contribute to setting priorities for the users' needs for flexible health services and enabling more patients to be treated near their homes.

If the study finds evidence of positive health gains for the individual people with diabetes and contributes to high quality of care, this new model can be implemented in the entire Stavanger Hospital Trust. This approach will enable the multidisciplinary team in specialist health care to be used more appropriately, and the team will be more accessible for health care personnel in municipal primary health care. This model can be transferred to other hospital trusts and contribute to improving knowledge on diabetes among nurses in municipal primary health care.

The main study confirmed that TM was non-inferior in traditional treatment with regard to healing time (primary outcome). The TM group had a signiﬁcantly lower proportion of amputations, and there were no signiﬁcant differences in the proportion of deaths, number of consultations, or patient satisfaction between groups, although the direction of the effect estimates for these clinical outcomes favored the TM group.

There is a need to continue the study with additional patients to gain more knowledge about the extent to which the telemedicine follow-up affects the number of consultations (secondary outcome), inclusion of participants during 2019-2021. In addition, there is a need for more knowledge about the effect of telemedicine follow-up for patients with leg ulcers and in people without diabetes. The investigators have used qualitative interview as a process evaluation in this study and will investigate process variables more systematically in the further follow-up. By examining how the services are organized (organization and structure) the investigators will gain knowledge how the variation in the organization of telemedicine follow-up is affecting the outcome.

ELIGIBILITY:
Inclusion Criteria:

* people with type 1 or type 2 diabetes with a new foot ulcer presenting for the first time within a period of 6 months and people without diabetes presenting a venous leg ulcer
* The participants must be able to read and speak Norwegian.
* The participants must be 20 years or older.

Exclusion Criteria:

- people treated for an diabetes foot ulcer on the ipsilateral foot during the past 6 months in specialist health care

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
healing time for leg ulcer and/or diabetes related foot ulcer | one year
  Healing time for leg ulcer and/or diabetes related foot ulcer measured from the time the person is included in the study until the foot ulcer is healed or the study ends (after 12 months). The effect will be measured in terms of hazard ratios (HR) and sub-hazard ratio (SHR) with healing as the endpoint and non-inferiority will be defined as <40% increased healing time in the TM-group, i.e. the lower 95% confidence limit should not be lower than 0.60.

SECONDARY OUTCOMES:
Total number of consultations per patient | one year
  Number of consultations from baseline until the foot ulcer has healed
sequela directly related to the foot ulcer | one year
  From baseline until the foot ulcer has healed sequelae directly related to the foot ulcer: infection, hospitalization, osteomyelitis and vascular surgery during the study
Diabetes-related stress | one year
  Diabetes-related stress, measured by using the Problem Areas in Diabetes. Measured at baseline and when the ulcer has healed (or the end of the study)
Symptoms of anxiety and depression | one year
  symptoms of anxiety and depression, measured by using the Hospital Anxiety and Depression Scale at baseline and the end of the study.
Nordic Patient Experiences Questionnaire | one year
  Patient satisfaction with health care, measured by using the Nordic Patient Experiences Questionnaire. Measured at baseline and the end of the study.
EQ-5D | one year
  Health status and cost utility, measured by using the EQ-5D from the EuroQol Group at baseline and the end of the study.
Sick leave | one year
  Sick leave (number of days with a medical certificate) measured by obtaining data from the Norwegian Sick Leave Registry measured from baseline unntil the ulcer is healed (or at the end of the study)
A new foot ulcer appears, the incidence of amputation and survival. | 2 and 3 years after the end of the study
  The time elapsing before a new foot ulcer appears, the incidence of amputation and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein M. Iversen, PhD, Principal Investigator — Helse Stavanger HF
Locations (3):
- Norway (3):
  - Stavanger HF, Stavanger, Rogaland
  - Haukeland University Hospital, Bergen
  - Stord Hospital, Helse Fonna HF, Leirvik

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blytt KM, Kolltveit BH, Graue M, Robberstad M, Ternowitz T, Carlsen S, Iversen MM. The implementation of telemedicine in wound care: a qualitative study of nurses' and patients' experiences. BMC Health Serv Res. 2024 Sep 29;24(1):1146. doi: 10.1186/s12913-024-11620-w. PMID 39343892
- [Derived] Iversen MM, Igland J, Smith-Strom H, Ostbye T, Tell GS, Skeie S, Cooper JG, Peyrot M, Graue M. Effect of a telemedicine intervention for diabetes-related foot ulcers on health, well-being and quality of life: secondary outcomes from a cluster randomized controlled trial (DiaFOTo). BMC Endocr Disord. 2020 Oct 21;20(1):157. doi: 10.1186/s12902-020-00637-x. PMID 33087074
- [Derived] Smith-Strom H, Igland J, Ostbye T, Tell GS, Hausken MF, Graue M, Skeie S, Cooper JG, Iversen MM. The Effect of Telemedicine Follow-up Care on Diabetes-Related Foot Ulcers: A Cluster-Randomized Controlled Noninferiority Trial. Diabetes Care. 2018 Jan;41(1):96-103. doi: 10.2337/dc17-1025. Epub 2017 Nov 29. PMID 29187423
- [Derived] Smith-Strom H, Iversen MM, Graue M, Skeie S, Kirkevold M. An integrated wound-care pathway, supported by telemedicine, and competent wound management-Essential in follow-up care of adults with diabetic foot ulcers. Int J Med Inform. 2016 Oct;94:59-66. doi: 10.1016/j.ijmedinf.2016.06.020. Epub 2016 Jun 29. PMID 27573312
- [Derived] Iversen MM, Espehaug B, Hausken MF, Graue M, Ostbye T, Skeie S, Cooper JG, Tell GS, Gunther BE, Dale H, Smith-Strom H, Kolltveit BC, Kirkevold M, Rokne B. Telemedicine Versus Standard Follow-Up Care for Diabetes-Related Foot Ulcers: Protocol for a Cluster Randomized Controlled Noninferiority Trial (DiaFOTo). JMIR Res Protoc. 2016 Jul 18;5(3):e148. doi: 10.2196/resprot.5646. PMID 27430301
- [Derived] Kolltveit BC, Gjengedal E, Graue M, Iversen MM, Thorne S, Kirkevold M. Telemedicine in diabetes foot care delivery: health care professionals' experience. BMC Health Serv Res. 2016 Apr 18;16:134. doi: 10.1186/s12913-016-1377-7. PMID 27091459